CLINICAL TRIAL: NCT04108793
Title: Effectiveness of Home-based Rehabilitation Program in Minimizing Disability and Secondary Falls After a Hip Fracture: A Randomized Controlled Trial
Brief Title: Effectiveness of Home-based Rehabilitation Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr. Shahryar Noordin, Associate Professor and orthopedic surgeon, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1533
Record Dates: First submitted 2019-09-24; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Fall

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study is an open label trial where patients, orthopedic surgeons, Nurses, and physical therapist will be aware of the intervention group. Therefore, no blinding or allocation concealment will be performed. However, the research assistant who will assess incidence of fall on telephone call will be kept blinded to ensure blinded data assessing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): The Intervention group will be given a program of progressive balance and lower limb strengthening exercises twice a week for 3 months. All exercises will include 5 minutes warm-up exercises. The lower limb extensor muscle groups (hip & knee extensors and ankle plantar flexors) will be targeted with exercises designed to enhance postural control (i.e. balance) and muscle strength. The balance exercises include standing with a decreased base of support, forwards and sideways stepping/walking, and graded reaching activities in standing. Strengthening exercises will include sit-to-stand, forward and lateral step-ups onto a small block, semi squats and heel raises in standing. Standard principles governing frequency, volume, duration, intensity and progression of exercise will be applied. Cueing strategies will be used to reduce freezing. T
  Interventions: Other: Physiotherapy exercises
- Control Arm (No Intervention): The control arm will receive the usual standard postoperative rehabilitation after a bipolar hemiarthroplasty/ total hip arthroplasty which will include in hospital rehabilitation and a maximum of 5 visits postoperatively

INTERVENTIONS:
Other: Physiotherapy exercises — The intervention group will receive an extended home-based rehabilitation program twice a week continued for 3 months (12 weeks) after discharge funded by the study.
  Arms: Intervention Arm

SUMMARY:
This study will be an open label, simple randomized controlled trial at a single hospital. The two arms will be equally allocated on a 1:1 ratio into intervention and control groups. The control arm will receive the usual standard postoperative rehabilitation after a bipolar hemiarthroplasty/ total hip arthroplasty which will include in hospital rehabilitation and a maximum of 5 visits postoperatively, arranged and funded by the patient as feasible. The intervention group will receive an extended home-based rehabilitation program twice a week continued for 3 months (12 weeks) after discharge funded by the study. The study will be conducted solely at Aga Khan University Hospital. The care providers involved with the study will include orthopaedic consultants, Family medicine physician, physiotherapist, and orthopaedic nurses. A total of 224 elderly patients aged 60 years and above undergoing hip fracture surgery will be evenly divided into intervention and control arms. The Primary outcome of the study is incidence of falls. Falls will be measured 3 monthly by research-assistant follow-up telephone calls for both the groups. Face to face interview which will be conducted in routine follow-up visits of all patients (both groups) will include assessment physical performance using Short Physical Performance Battery (SPPB) tool.

DETAILED DESCRIPTION:
Hip fractures are a major health problem globally and are associated with increased morbidity, mortality, and substantial economic costs. Successful operative treatment of hip fracture patients is necessary for the optimization of post-op mobility and functional recovery of the patient. Rehabilitation after surgical stabilization of a hip fracture is crucial in order to restore pre-fracture function and to avoid long-term institutionalization. The probability of long-term confinement can be as high as 25% if the fracture is not fixed.

The combination of high incidence of fall and a high susceptibility to injury is a major public health concern among elderly population. This propensity for fall-related injury in elderly persons stems from a high prevalence of co morbid diseases such as osteoporosis and age-related physiological decline (e.g. slower reflexes) that make even a relatively mild fall, potentially dangerous The development and implementation of effective strategies to minimize disability and falls among older people is an urgent public health challenge due to the increasing proportion of older people in the global population. Besides, for many individuals, the risk of falls and disability after hospital discharge decreases with time. However, for a significant proportion, this is not the case. Many patients after discharge are readmitted with second fracture to the hospitals due to lack of acute rehabilitation programs. Therefore, we have designed a post-discharge home-based physical rehabilitation intervention program to minimize disability and falls in this high-risk elderly population.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 60 years
2. able to walk independently with or without a walking frame prior to the fracture
3. diagnosis of proximal femoral fracture
4. history of fall
5. surgical procedure Bipolar hemiarthroplasty / total hip replacement and postoperative ambulatory status weight bearing as tolerated.

Exclusion Criteria:

1. unable to walk more than one meter despite assistance with a walking aid
2. legally blind
3. progressive neurological disease (e.g. Parkinson's disease, dementia)
4. Any medical condition precluding exercise (e.g. unstable cardiac disease) or other uncontrolled chronic conditions that would interfere with the safety and conduct of the training and testing protocol or interpretation of results.
5. Patients undergoing dynamic hip screw (DHS)

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
occurrence of secondary fall. | All the Patients (both groups) will be contacted after every 3 months for the period of two years via telephone call to assess occurrence of fall
  The Primary outcome of the study is occurrence secondary fall. Follow-ups will be done 3 monthly by research-assistant using telephone calls for both the groups to assess if occurrence of secondary fall. A fall will be defined according to the Kellogg definition as an incident in which the body unintentionally comes to rest on the ground or other lower level which is not as a result of a violent blow, loss of consciousness, and sudden onset of paralysis as in a stroke or an epileptic seizure.
  Falls will be assessed by comparing the number of falls in intervention and control groups. The occurrence of fall in each group will also be compared.

SECONDARY OUTCOMES:
Physical Mobility and Mobility-related disability | the performance-based mobility measure will be marked at every routine follow-up for up to two years using face to face interview to assess the overall trend.
  The performance-based mobility measure will be the lower extremity Summary Performance Score version of the Short Physical Performance Battery (SPPB). This battery gives a composite score based on timed performance of three mobility tasks: the ability to stand up for up to 10 seconds with feet in different positions (together side by side, semi-tandem and tandem), 4-meter walk and time to rise from a chair 5 times. The short performance based mobility tool is a valid and reliable tool with test retest validity ranging from 0.83 to 0.89

CONTACTS AND LOCATIONS:
Overall Officials: Shahryar Noordin, MBBS,FCPS, Principal Investigator — Aga Khan University

IPD SHARING:
Plan to Share IPD: Yes
Manuscripts, conferences, symposiums
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After October 2021
Access Criteria: Contact to PI

REFERENCES:
- [Derived] Fairhall NJ, Dyer SM, Mak JC, Diong J, Kwok WS, Sherrington C. Interventions for improving mobility after hip fracture surgery in adults. Cochrane Database Syst Rev. 2022 Sep 7;9(9):CD001704. doi: 10.1002/14651858.CD001704.pub5. PMID 36070134
- [Derived] Sadruddin Pidani A, Sabzwari S, Ahmad K, Mohammed A, Noordin S. Effectiveness of home-based rehabilitation program in minimizing disability and secondary falls after a hip fracture: Protocol for a randomized controlled trial. Int J Surg Protoc. 2020 Jun 18;22:24-28. doi: 10.1016/j.isjp.2020.06.002. eCollection 2020. PMID 32695954